CLINICAL TRIAL: NCT05453422
Title: The Effect of Self-Acupressure on Pain, Fatigue and Sleep Quality in Patients With Systemic Lupus Erythematosus: A Randomized Controlled Study
Brief Title: Self-Acupressure on Pain, Fatigue and Sleep Quality in Systemic Lupus Erythematosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, Director, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 8990
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Sleep Disorder
Keywords: Fatigue; Pain; Sleep quality; Systematic lupus erythemasus
MeSH Terms: conditions — Sleep Wake Disorders; Fatigue; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Masking Description: Self-Acupressure and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Acupressure (Experimental): Each application to the acupressure points (H17, L14, ST36, SP6) will be done in 2 minutes and right and left)
  Interventions: Other: Self-Acupressure
- Control group (No Intervention): Routine maintenance will be applied.

INTERVENTIONS:
Other: Self-Acupressure — Acupressure is a therapy method performed with an instrument or hand, fingertip, palm, elbow, knee, thumb relaxation and wrist bands on various points representing the waist organs in order to ensure the continuation and balance of the energy in our body.
  Arms: Self-Acupressure

SUMMARY:
The aim of this study is to examine the effect of Self-acupressure application on pain, fatigue and sleep quality in sle patients.

DETAILED DESCRIPTION:
Acupressure is a therapy method performed with an instrument or hand, fingertip, palm, elbow, knee, thumb relaxation and wrist bands on various points representing the waist organs in our body in order to ensure the continuation and balance of the energy in our body.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18,
* Not using acupressure and similar integrative treatment methods,
* Not having a verbal communication disability (hearing and speaking),
* Not having a diagnosed psychiatric disorder,
* Not having a cognitive problem,
* Getting a score between 1-10 on the Piper Fatigue Scale,
* Getting a score between 1-10 on the VAS pain scale
* Agree to participate in the research.
* Not being in the active period of SLE (exacerbation in the last 3 months or not using steroids for 3 months)
* Not using other complementary and integrated health practices in the treatment process

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | At the end of Sessions 1 (each Session 2 days a week).
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
Visual Analog Scale | At the end of Sessions 16 (each Session 2 days a week).
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
The Piper Fatigue Scale | At the end of Sessions 1 (each Session 2 days a week).
  The Piper Fatigue Scale is a 22-item, self-reported scale. A total score of fatigue was recorded.
The Piper Fatigue Scale | At the end of Sessions 16 (each Session 2 days a week).
  The Piper Fatigue Scale is a 22-item, self-reported scale. A total score of fatigue was recorded.
The Richards-Campbell Sleep Questionnaire | At the end of Sessions 1 (each Session 2 days a week).
  This brief five-item questionnaire was used to evaluate perceived sleep depth, sleep latency (time to fall asleep), number of awakenings, efficiency (percentage of time awake), and sleep quality. It also includes a sixth item evaluating perceived night-time noise. Each item is evaluated on a scale of 0-100 with a visual analogue scale technique. A score of 0-25 indicates very poor quality sleep, whereas a score of 76-100 indicates very good sleep quality.
The Richards-Campbell Sleep Questionnaire | At the end of Sessions 16 (each Session 2 days a week).
  This brief five-item questionnaire was used to evaluate perceived sleep depth, sleep latency (time to fall asleep), number of awakenings, efficiency (percentage of time awake), and sleep quality. It also includes a sixth item evaluating perceived night-time noise. Each item is evaluated on a scale of 0-100 with a visual analogue scale technique. A score of 0-25 indicates very poor quality sleep, whereas a score of 76-100 indicates very good sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz Özer, PhD, Study Director — Istanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aranow C, Atish-Fregoso Y, Lesser M, Mackay M, Anderson E, Chavan S, Zanos TP, Datta-Chaudhuri T, Bouton C, Tracey KJ, Diamond B. Transcutaneous auricular vagus nerve stimulation reduces pain and fatigue in patients with systemic lupus erythematosus: a randomised, double-blind, sham-controlled pilot trial. Ann Rheum Dis. 2021 Feb;80(2):203-208. doi: 10.1136/annrheumdis-2020-217872. Epub 2020 Nov 3. PMID 33144299
- [Result] Wang T, Zhang Q, Xue X, Yeung A. A systematic review of acupuncture and moxibustion treatment for chronic fatigue syndrome in China. Am J Chin Med. 2008;36(1):1-24. doi: 10.1142/S0192415X08005540. PMID 18306446